CLINICAL TRIAL: NCT00460343
Title: Implementation of a Pharmacy-Intervention to Establish and if Necessary Improve Adherence to Antihypertensive Therapy. A Cluster Randomized Trial.
Brief Title: Pharmacy Implementation Trial: Adherence to Antihypertensive Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Zorgverzekeraar CZ (Other); Scientific Institute for Dutch Pharmacists, The Netherlands (Other)
Responsible Party: Caroline van de Steeg-van Gompel, Scientific Institute for Quality of Healthcare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: WOK/WINAp/CZ-03; CMO-nr 2006/072
Record Dates: First submitted 2007-04-04; First posted 2007-04-13 (Estimated); Last update posted 2008-07-10 (Estimated); Status verified 2008-07

CONDITIONS: Hypertension
Keywords: patient non-adherence; antihypertensive agents; community pharmacy services; professional roles
MeSH Terms: conditions — Hypertension; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- max (Experimental)
  Interventions: Other: extensive implementation programme
- min (Active Comparator)
  Interventions: Other: control

INTERVENTIONS:
Other: extensive implementation programme — experimental pharmacists follow an extensive implementation programme. They attend two interactive half a day educational meetings tailored to individual needs: one at start of the intervention, and one in May or September 2007. Special attention is given to multiprofessional cooperation with general practitioners and nurse practitioners. Additionally, guided by their own project planning pharmacists receive three or more telephone calls, both as a reminder, feedback, and in order to investigate whether they need any more help.
  Arms: max
Other: control — pharmacists only receive a written manual with instructions to implement the patient compliance intervention.
  Arms: min

SUMMARY:
The purpose of this study is to determine the effectiveness of maximal support of community pharmacies to implement a pharmaceutical care model for establishing and - if necessary - improving adherence to antihypertensive medication in patients with medication-resistant hypertension.

DETAILED DESCRIPTION:
Cardiovascular disease is the main cause of death in large parts of the world. Hypertension is an important risk factor for cardiovascular disease. Although hypertension treatment has improved in the last decade, the effectiveness of antihypertensive therapy still needs attention. Adherence to medication appears to play an important role in that.

Pharmacists can support the general practitioners in their efforts to optimize antihypertensive therapy, by establishing adherence to medication of patients with hypertension in spite of the use of one or more antihypertensive drugs. This is performed with the electronic Medication Event Monitoring System (MEMS®). Registered adherence and accompanying blood pressure are discussed with the patient by the GP.

Implementation of the above-mentioned intervention is studied in two randomized groups of pharmacies. One group receives minimal support in the intervention, the other group also receives interactive educational meetings, reminders and feedback, and support of multiprofessional cooperation.

ELIGIBILITY:
Inclusion Criteria:

* pharmacies: resident in the south of the Netherlands
* patients:

  * 18 years or older
  * diagnosis of hypertension
  * systolic blood pressure between 150 and 180 mm Hg despite the use of antihypertensive drug(s)
  * indication for treatment escalation

Exclusion Criteria:

* patients:

  * impossibility to establish blood pressure properly
  * patient treated by medical specialist
  * change of antihypertensive therapy because of adverse effects of current medication
  * insisting on using dose organisers
  * not managing their drug intake themselves
  * not able to come to the pharmacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
the number of patients included for intervention | 9 months after start of the study

SECONDARY OUTCOMES:
improvement of systolic blood pressure | 2 and 5 months after inclusion
treatment escalation of patients after inclusion into the study | 5 months after inclusion
the percentage of GP's in PTAM that cooperates in the intervention | 9 months after start of the study

CONTACTS AND LOCATIONS:
Overall Officials: Peter G de Smet, PhD, Principal Investigator — Radboud University Medical Center; Michel Wensing, PhD, Study Director — Scientific Institute for Quality of Healthcare

REFERENCES:
- [Background] Ragot S, Sosner P, Bouche G, Guillemain J, Herpin D. Appraisal of the knowledge of hypertensive patients and assessment of the role of the pharmacists in the management of hypertension: results of a regional survey. J Hum Hypertens. 2005 Jul;19(7):577-84. doi: 10.1038/sj.jhh.1001859. PMID 15830000
- [Background] Krousel-Wood M, Thomas S, Muntner P, Morisky D. Medication adherence: a key factor in achieving blood pressure control and good clinical outcomes in hypertensive patients. Curr Opin Cardiol. 2004 Jul;19(4):357-62. doi: 10.1097/01.hco.0000126978.03828.9e. PMID 15218396
- [Background] Lee JK, Grace KA, Taylor AJ. Effect of a pharmacy care program on medication adherence and persistence, blood pressure, and low-density lipoprotein cholesterol: a randomized controlled trial. JAMA. 2006 Dec 6;296(21):2563-71. doi: 10.1001/jama.296.21.joc60162. Epub 2006 Nov 13. PMID 17101639
- [Background] Burnier M, Schneider MP, Chiolero A, Stubi CL, Brunner HR. Electronic compliance monitoring in resistant hypertension: the basis for rational therapeutic decisions. J Hypertens. 2001 Feb;19(2):335-41. doi: 10.1097/00004872-200102000-00022. PMID 11212978
- [Background] Waeber B, Vetter W, Darioli R, Keller U, Brunner HR. Improved blood pressure control by monitoring compliance with antihypertensive therapy. Int J Clin Pract. 1999 Jan-Feb;53(1):37-8. PMID 10344064
- [Background] Carter BL, Zillich AJ, Elliott WJ. How pharmacists can assist physicians with controlling blood pressure. J Clin Hypertens (Greenwich). 2003 Jan-Feb;5(1):31-7. doi: 10.1111/j.1524-6175.2003.01460.x. PMID 12556651
- [Background] Fahey T, Schroeder K, Ebrahim S. Interventions used to improve control of blood pressure in patients with hypertension. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD005182. doi: 10.1002/14651858.CD005182. PMID 15654709
- [Background] Wetzels GE, Nelemans PJ, Schouten JS, Dirksen CD, van der Weijden T, Stoffers HE, Janknegt R, de Leeuw PW, Prins MH. Electronic monitoring of adherence as a tool to improve blood pressure control. A randomized controlled trial. Am J Hypertens. 2007 Feb;20(2):119-25. doi: 10.1016/j.amjhyper.2006.07.018. PMID 17261454